CLINICAL TRIAL: NCT06337266
Title: A Novel Online Calculator to Predict Long-term Survival and Recurrence Risk of Patients With Gastric Adenocarcinoma After Radical Gastrectomy : A Multicenter Real-world Study
Brief Title: A Novel Online Calculator to Predict Long-term Survival and Recurrence Risk of Patients With Gastric Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: 2024KY246
Record Dates: First submitted 2024-03-19; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: oxidative stress; inflammation; Gastric adenocarcinoma; nomogram; recurrence risk
MeSH Terms: conditions — Stomach Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Cohort

SUMMARY:
This study aimed to develop a novel Prognostic Oxidative Stress-Immune-Inflammatory Score (POSII Score) and introduce an innovative online calculator designed to predict long-term survival and assess the recurrence risk of gastric cancer (GC).

DETAILED DESCRIPTION:
From 2009 to 2020, this study analyzed GC patients underwent Radical Gastrectomy at three hospitals, dividing them into training, internal, and external validation cohorts. Twelve blood indicators were analyzed. The POSII Score was developed in the training cohort using the Least Absolute Shrinkage and Selection Operator (LASSO) technique. Additionally, two online nomogram calculators were created based on multivariate Cox regression within the training cohort and subsequently validated in internal and external validation cohorts.

ELIGIBILITY:
Inclusion Criteria:1) histopathologically diagnosed gastric adenocarcinoma, 2) undergoing radical gastrectomy for GC, 3) absence of tumor invasion into adjacent organs or distant metastasis, and 4) availability of complete laboratory data.

Exclusion Criteria: 1) non-adenocarcinoma gastric cancers, 2) gastric stump cancer, 3) receipt of neoadjuvant therapy, 4) a history of other malignancies, and 5) insufficient clinical data or follow-up information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a multicenter, retrospective cohort investigation involving GC patients who underwent radical gastrectomy at the Fujian Medical University Union Hospital (FMUUH), the First Affiliated Hospital of Gannan Medical University (FAHGMU) and Quzhou Affiliated Hospital of Wenzhou Medical University (QAHWMU) between January 2009 and June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3622 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
5-year OS | 5 years or 60 months
  overall survival, death, survival with tumor, deletion
5-year DFS | 5 years or 60 months
  Disease-free survival,Recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, M.D., Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No